CLINICAL TRIAL: NCT06924996
Title: Efficacy and Safety of Endovascular Thrombectomy in Acute Ischemic Stroke With Posterior Circulation Large Infarct: A Multicenter, Prospective, Cohort Study
Brief Title: Efficacy and Safety of Endovascular Thrombectomy in Acute Ischemic Stroke With Posterior Circulation Large Infarct
Status: Enrolling by invitation | Type: Observational
Sponsor: Feng Gao (Other)
Responsible Party: Sponsor-Investigator, Feng Gao, Interventional Neuroradiology, Department of Neurology, Beijing Tiantan Hospital, Capital Medical University
Organization: Capital Medical University (Other)
Other Study IDs: KY2023-106-02
Record Dates: First submitted 2025-04-10; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Acute Basilar Artery Occlusion; Posterior Circulation Large Infarct

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endovascular Thrombectomy (EVT): The EVT group would include the following interventions: stent-retriever thrombectomy, aspiration thrombectomy, balloon angioplasty and/or stenting, intra-arterial medication administration, or a combination of these approaches.
  Interventions: Procedure: Endovascular Thrombectomy (EVT)
- Best Medical Management (BMM): BMM was tailored according to institutional guidelines and included intravenous thrombolysis (IVT), antiplatelet therapy, anticoagulation, or multimodal combinations.

INTERVENTIONS:
Procedure: Endovascular Thrombectomy (EVT) — A maximum of six attempts to retrieve the thrombus in a single vessel can be made with any Solitaire AB/FR device or aspiration. In case an atherosclerotic lesion is found underlying the occlusive lesion, angioplasty and subsequent stenting through detachment of the Solitaire device will be allowed
  Groups: Endovascular Thrombectomy (EVT)

SUMMARY:
The purpose of this study is to evaluate whether endovascular thrombectomy (EVT) combined with best medical management (BMM) leads to better functional outcomes than BMM alone in patients with acute basilar artery occlusion with posterior circulation large infarct.

DETAILED DESCRIPTION:
This study is a multicenter, prospective, cohort study that prospectively enrolled consecutive patients with acute basilar artery occlusion and large core infarction in the posterior circulation, confirmed by imaging (CTA/MRA/DSA). Written informed consent was obtained from all participants or their legal representatives prior to enrollment. Patients were divided into the best medical management (BMM) group and the endovascular thrombectomy (EVT) group according to the treatment they received. This study adhered to the Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years old;
2. Acute ischemic stroke in the posterior circulation, the onset of stroke (or last well known) to the enrollment time within 24 hours;
3. CTA/MRA/DSA confirmed acute basilar artery occlusion;
4. Posterior circulation large infarct: NCCT or DWI showed pc-ASPECTS ≤ 5 points, or pontine midbrain index (PMI) ≥ 3 points;
5. NIHSS score ≥10 points after the onset of the stroke and before enrollment;
6. Able to live independently before the onset of the disease (mRS score ≤2 points);
7. The subject or legal representative is able to sign the informed consent form.

Exclusion Criteria:

1. Intracranial hemorrhage (except microhemorrhage) on CT/MRI ;
2. CT/MRI revealed large infarction in the cerebellar hemisphere, with significant mass effect causing compression of the fourth ventricle or brainstem;
3. CT or MRI showed bilateral complete thalamic infarction;
4. Occlusion of anterior and posterior circulation arteries confirmed by CTA/MRA/DSA;
5. The presence of intracranial tumors (except for small meningiomas and cerebral aneurysms with a diameter of <3mm);
6. Patients with known or highly suspected chronic basilar artery occlusion.;
7. Known severe allergy to contrast agents (except for mild rash);
8. Refractory hypertension (defined as systolic blood pressure > 185 mmHg or diastolic blood pressure >110 mmHg) that cannot be controlled by drug therapy;
9. Known pregnant or lactating females, or positive pregnancy test before enrollment;
10. Acute cerebral infarction within 48 hours after cardiovascular and cerebrovascular intervention or major surgery (patients more than 48 hours can be enrolled).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute basilar artery occlusion with large infarct
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of modified Rankin scale 0-3 at 90 (±14) days after enrollment | 90 (±14) days
  The modified Rankin scale (mRS) ranged from 0 to 6, with a score of 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but remaining able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death.

SECONDARY OUTCOMES:
Ordinal Shift analysis of mRS score at 90 (±14) days after enrollment | 90 (±14) days
  The modified Rankin scale (mRS) ranged from 0 to 6, with a score of 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but remaining able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death.
Rate of mRS 0-2 at 90 (±14) days after enrollment | 90 (±14) days
  The modified Rankin scale (mRS) ranged from 0 to 6, with a score of 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but remaining able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death.
Rate of Functional health status and quality of life (EuroQol Five Dimensions) at 90 (±14) days after enrollment | 90 (±14) days
  EuroQol Five Dimensions (EQ-5D) is a standardized instrument for measuring the general health status. Rated level can be coded as a number 1, 2, 3, 4 or 5, which indicates having no problems for 1, having some problems for 2, having moderate problems for 3, having serious problems for 4 and having extreme problems for 5

OTHER OUTCOMES:
Mortality within 90 (±14) days | 90 (±14) days
  all-cause mortality
Rate of Symptomatic intracranial hemorrhage (SICH) | 24-72 hours
  Symptomatic intracranial hemorrhage (SICH) within 24-72 hours after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: gao feng, professor, Study Chair — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China